CLINICAL TRIAL: NCT01126996
Title: An Observational Study Into the Maintenance of Seroprotection Against Meningococcal Serogroup C Disease Throughout Childhood Following a Single Dose of a Conjugated Meningococcal Serogroup C Vaccine Administered to Toddlers
Brief Title: Understanding the Persistence of Immunity After MenC Vaccines
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Ms Heather House, University of Oxford, CTRG
Other Study IDs: OVG 2009/06
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: MenC conjugate vaccine; Healthy children previously vaccinated against MenC
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MenC vaccinated healthy children: Children who received a single dose of a MenC conjugate vaccine at age 1-3 years 10 years earlier.
  Interventions: Procedure: Venepuncture

INTERVENTIONS:
Procedure: Venepuncture — 1. Venepuncture and blood sample collection in 2010 in a sample of children who received a single dose of a MenC conjugate vaccine at age 1-3 years 10 years earlier.
  2. A booster dose of a MenC conjugate vaccine (optional).

SUMMARY:
Neisseria meningitidis occurs worldwide as endemic disease1 and is a major cause of invasive infections such as meningitis and septicaemia. Three protein-polysaccharide conjugate serogroup C meningococcal (MenC) vaccines were developed in the late 1990's and an accelerated programme of clinical trials in the UK led to licensure of these MenC vaccines in 1999 and these vaccines were introduced into the routine infant immunisation schedule at 2, 3 and 4 months. However, children who were aged 1-18 years in 2000 only received a single dose of a MenC conjugate vaccine during the mass immunisation campaign.

Previous studies have demonstrated rapid waning of MenC specific antibody concentrations and serum bactericidal antibody (SBA) titres following immunisation in young children. A cross-sectional review on rates of sero-protection against MenC disease in the UK has demonstrated that the majority of children who were immunised with a single dose of a MenC conjugate vaccine between the ages of 1-10 did not have protective titres of MenC SBA 7 years after the immunisation campaign. As this cohort of children reaches adolescence there is a risk of increased transmission of the organism and a resurgence of meningococcal disease in children who do not have protective levels of antibody. There is thus a need to conduct a study evaluating the changes in MenC SBA titres over time in children who received a single dose of a MenC vaccine in early childhood which is the main objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant whose parent is willing and able to give informed consent for participation in the study.
* Participant who gives assent for participation in the study.
* Male or Female, aged 11 to 13 years.
* Known to be free from medical problems as determined by a medical history and clinical assessment
* Participated in the University of Oxford clinical trial: U01-Td5I-303/ C01.183

Exclusion Criteria:

* History of invasive meningococcal C disease
* Any vaccination against MenC disease with the exception of a single dose in 2000 during the nationwide MenC immunisation campaign
* Confirmed or suspected immunosuppressive or immunodeficient conditions, including human immunodeficiency virus (HIV) infection.
* Major congenital defects or serious chronic illness

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children who participated in the U01-Td5I-303/ C01.183 study from 2001 to 2007 who will be aged 11 to 13 years in 2010, all of whom would have received a single dose of a MenC conjugate vaccine in 2000 as part of the nationwide immunisation campaign.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with rSBA titres >1:8 (correlate of protection) | 6 months

SECONDARY OUTCOMES:
MenC rSBA GMTs at all time points when sera is available after receiving a dose of MenC vaccine | 6 months
Percentage of children at each time point with MenC SBA titres >1:8 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Snape, Principal Investigator — University of Oxford
Locations (1):
- Oxford Vaccine Group, University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Background] Khatami A, Peters A, Robinson H, Williams N, Thompson A, Findlow H, Pollard AJ, Snape MD. Maintenance of immune response throughout childhood following serogroup C meningococcal conjugate vaccination in early childhood. Clin Vaccine Immunol. 2011 Dec;18(12):2038-42. doi: 10.1128/CVI.05354-11. Epub 2011 Oct 28. PMID 22038849